CLINICAL TRIAL: NCT04394013
Title: A Web-Based Gentle Body Stretching to Alleviate Loneliness and Improve Mental Fitness During COVID-19 Isolation Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Teoh Siew Li, Lecturer, Monash University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 180320201
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Arm (Experimental): The content of the approximately 20 minutes video is recorded in advance of the intervention by a certified teacher with teaching experience. The 20 minutes session consists of a series of body stretching exercises (around 17 different gentle and simple stretches from head to toe) with the incorporation of breathing technique (i.e. when to breathe in and breathe out). The whole body stretching exercise is performed with a sitting position, ideally on an exercise mat. As mentioned above, the participants are required to conduct the stretching exercise by following the guidance video for at least 5 days weekly for at least 2 weeks duration. The video will be uploaded onto a webpage which requires participants to log in and view the video. The webpage and video will be accessible through computers and mobile phones.
  Interventions: Behavioral: Mindfulness intervention
- Non-mindfulness Arm (Active Comparator): In this study, for control group, the participants are instructed with a similar video content as the intervention group, minus the incorporation of breathing technique, as breathing technique is hypothesised to be a key component of mindfulness.
  Interventions: Behavioral: Non-Mindfulness intervention

INTERVENTIONS:
Behavioral: Mindfulness intervention — Gentle body stretching with the incorporation of breathing technique
  Arms: Mindfulness Arm
Behavioral: Non-Mindfulness intervention — Gentle body stretching without the incorporation of breathing technique
  Arms: Non-mindfulness Arm

SUMMARY:
During the COVID-19 pandemic, individuals are having to stay at home in quarantine to reduce the risk of transmission of the virus. Depending on the number of occupants and the dwelling space available, this can lead to household crowding, which can have an effect on mental health. In addition, the closing of leisure facilities, including restaurants, cafes and, with the need to self-isolate and socially distance, has led to loneliness. The focus on "loneliness" has recently been on a rise, and being described as an epidemic, especially when it has been shown to be associated with various diseases as well as increased risk of mortality. Studies conducted on participants in isolation has shown increased mental health issues including anxiety, stress and depression.

Mindfulness intervention has been shown to alleviate mental health issues including loneliness. However, to date, there is limited studies examining the effectiveness of a remote mindfulness intervention. This proposal aims to deliver a remote mindfulness program that can be accessible by participants easily and even during the isolation period. This intervention will investigate the effectiveness and safety in elevating mental health issues faced by the general population.

DETAILED DESCRIPTION:
Loneliness, mindfulness and quality of life will be assessed as the primary outcome of the study. A mindfulness video will be used as the intervention for participants, and is compared with a group with similar video content without mindfulness component. The effect of changes in primary outcome will be assessed between groups after 2-4weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Loneliness (UCLA-8 Loneliness Scale) | 2-4weeks
  Measured using University of California, Los Angeles (UCLA)-8 Loneliness Scale; Higher score indicates higher loneliness level
Mindfulness (FFMQ) | 2-4weeks
  Five-Facet Mindfulness Questionnaire (FFMQ); Higher score indicates higher mindfulness level
Quality of life (EQ-5D-5L Questionnaire) | 2-4weeks
  EQ-5D-5L Questionnaire; Higher score indicates higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Siew Li Teoh, PhD, Principal Investigator — Monash University Malaysia
Locations (1):
- Monash University Malaysia, Subang Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Upon request via direct contact to researcher

REFERENCES:
- [Derived] Jong FJX, Lee CCW, Ting RS, Lin MH, Ong LK, Quek XF, Lee SWH, Ng ALO, Teoh SL. Effects of online mindful stretching exercises for loneliness, mindfulness, and hair cortisol: A mixed method study. Explore (NY). 2025 Jul-Aug;21(4):103204. doi: 10.1016/j.explore.2025.103204. Epub 2025 Jun 26. PMID 40614537